CLINICAL TRIAL: NCT01661322
Title: Safety and Efficacy of Intensive Versus Guideline Antiplatelet Therapy in High Risk Patients With Recent Ischaemic Stroke or Transient Ischaemic Attack: a Randomised Controlled Trial
Brief Title: Triple Antiplatelets for Reducing Dependency After Ischaemic Stroke
Acronym: TARDIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial reached a definitive answer ahead of full recruitment.
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08093; 2007-006749-42 (EudraCT Number)
Record Dates: First submitted 2012-07-23; First posted 2012-08-09 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Stroke
Keywords: Acute ischaemic stroke; TIA
MeSH Terms: conditions — Stroke | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive antiplatelet therapy (Active Comparator): Participants in the intensive antiplatelet group will receive Aspirin+Dipyridamole+Clopidogrel triple therapy for 28-30 days (to cover the period of maximum risk of recurrence) along with standard 'best care' (including lifestyle advice, BP and lipid lowering). Clop will be given as a loading dose of 300 mg,12 then 75 mg daily, Asp as a loading dose of 300 mg,22 then 75 mg daily, and Dip modified release 200 mg twice daily 9 for 28-30 days.
  Interventions: Drug: Aspirin, Dipyradimole, Clopidogrel
- Guideline antiplatelet therapy (No Intervention): This may be one or two antiplatelet drugs, as per standard treatment. Clopidogrel or aspirin and dipyridamole.

INTERVENTIONS:
Drug: Aspirin, Dipyradimole, Clopidogrel — Participants in the intensive antiplatelet group will receive Asp+Dip+Clop triple therapy for 28-30 days (to cover the period of maximum risk of recurrence) along with standard 'best care' (including lifestyle advice, BP and lipid lowering). Clop will be given as a loading dose of 300 mg,12 then 75 mg daily, Asp as a loading dose of 300 mg,22 then 75 mg daily, and Dip modified release 200 mg twice daily 9 for 28-30 days.
  Other Names: Aspirin; Dipyradimole; Clopidogrel
  Arms: Intensive antiplatelet therapy

SUMMARY:
The risk of recurrence is greatest immediately after stroke or Transient Ischaemic Attack (TIA). Existing prevention strategies (antithrombotic, lipid/blood pressure lowering, endarterectomy) reduce, not abolish, further events. Dual antiplatelet therapy - aspirin & clopidogrel (AC) for IHD, aspirin & dipyridamole (AD) for stroke, is superior to aspirin monotherapy. The investigators hypothesise that triple antiplatelet therapy (ACD) will be superior to AD in patients at high-risk of recurrence, providing bleeding does not become excessive.

Design: TARDIS is a multicentre, parallel-group, prospective, randomised, open-label, blinded-endpoint, controlled trial. In the start-up phase, the investigators will assess over 3 years the safety, tolerability and feasibility of intensive therapy (ACD) versus guideline therapy (AD) given for 1 month in 750 patients with acute stroke/TIA. The main phase will then assess the safety and efficacy of ACD in up to 3500 patients. The primary outcome is ordinal stroke (fatal/severe non-fatal/mild/TIA/none) at 90 days. Secondary outcomes include death, MI, vascular events, function, bleeding, serious adverse events; sub-studies will assess cerebral emboli and platelet function.

DETAILED DESCRIPTION:
2.1 Purpose To perform a randomised trial assessing the efficacy, safety and tolerability of intensive antiplatelet therapy (Asp+Dip+Clop) versus guideline antiplatelet therapy (Asp+Dip or Clop) in patients with recent ischaemic stroke or TIA and who are at high risk of recurrence.

2.2 Primary Objective To assess ordinal stroke severity at 90 days after short-term administration (1 month) of intensive antiplatelet therapy versus guideline therapy in patients with very recent ischaemic stroke or TIA.

2.3 Secondary Objectives

1. To assess the safety of short-term administration (1 month) of intensive antiplatelet therapy versus guideline therapy in patients with very recent ischaemic stroke or TIA.
2. To further assess, in high risk patients with stroke/TIA, whether:

ii. it is feasible to administer intensive therapy acutely and is tolerable to take for 1 month, iii. intensive therapy is superior in respect of surrogate markers such as platelet function.

iv. intensive therapy improves functional outcome

ELIGIBILITY:
Inclusion Criteria:

Adults at high risk of recurrent ischaemic stroke:

1. Age ≥ 50 years
2. Within 48 hours of ictus (24-48 hours if thrombolysed)
3. TIA with limb weakness and/or dysphasia lasting between 10 minutes and < 24 hours with no residual symptoms and presenting with any of the following

   * ABCD2 score > 4, or
   * Crescendo TIA or
   * Already on dual antiplatelet therapy

   Note: Neuroimaging is not necessary for transient ischaemic attack. Crescendo TIA is > 1 TIA in one week and the onset time of last TIA is taken as time of ictus.
4. Ischaemic non cardioembolic stroke presenting with any of the following

   * Ongoing limb weakness and/or dysphasia of more than one hour duration
   * Resolved limb weakness of more than one hour duration with ongoing facial weakness
   * Ongoing isolated hemianopia of more than 1 hour duration with positive neuroimaging evidence to support the index event (e.g. ischaemic stroke in occipital lobe)
   * Resolved limb weakness and/or dysphasia between 24-48 hours after index event onset

   Note: Neuroimaging is essential for ischaemic stroke to exclude intracranial haemorrhage and/or non stroke diagnosis
5. Informed consent from participant. If the participant is unable to give meaningful consent e.g. due to dysphasia, confusion, or reduced conscious level, proxy consent may be obtained from a relative, carer or legal representative.

Exclusion Criteria:

1. Age < 50
2. Isolated sensory symptoms or vertigo/dizziness or facial weakness
3. Isolated hemianopia without positive neuroimaging evidence
4. Intracranial haemorrhage
5. Baseline neuroimaging showing parenchymal haemorrhagic transformation (PH I/II) of infarct, subarachnoid haemorrhage or other non ischaemic cause for symptoms
6. Presumed cardioembolic stroke (e.g. history or current AF, myocardial infarction within 3 months)
7. Participants with contraindications to, or intolerance of, aspirin, clopidogrel or dipyridamole.
8. Participants with definite need for treatment with aspirin, clopidogrel or dipyridamole individually or in combination (e.g. aspirin and clopidogrel for recent MI/acute coronary syndrome)
9. Participant has taken clopidogrel or dipyridamole after the index event but prior to randomisation (aspirin is allowed between ictus onset and randomisation)
10. Definite need for full dose oral (e.g. warfarin, dabigatran) or medium to high dose parenteral (e.g. heparin) anti-coagulation. NB Low dose heparin for DVT prophylaxis is allowed
11. Definite need for glycoprotein IIb-IIIa inhibitors
12. Received thrombolysis within the last 24 hours
13. No enteral access
14. Pre-morbid dependency (mRS > 2).
15. Severe high BP (BP > 185/110 mmHg).
16. Haemoglobin less than 10g/dL
17. Platelet count more than 600 x 109 /L or less than 100 x 109 /L
18. White cell count more than 30 x 109 /L or less than 3.5 x 109 /L
19. Major bleeding within 1 year (e.g. peptic ulcer, intracerebral haemorrhage).
20. Planned surgery during 3 month follow-up (e.g. carotid endarterectomy)
21. Concomitant STEMI or NSTEMI.
22. Stroke secondary to a procedure (e.g. carotid or coronary intervention)
23. Coma (GCS < 8)
24. Non-stroke life expectancy < 6 months
25. Dementia
26. Participation in another drug or devices trial concurrently or within 30 days. (participants may take part in observational studies or non-drug or devices trials)
27. Geographical or other factors that may interfere with follow-up e.g. no fixed address or telephone contact number, not registered with a GP, or overseas visitor.
28. Females of childbearing potential, pregnancy or breastfeeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3096 (Actual)
Dates: Start 2009-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome is ordinal stroke severity at 90 days | 90 days
  5-level ordinal stroke and TIA scale with stroke ordered by its severity using the modified Rankin Scale (mRS): fatal stroke / severe non-fatal stroke (mRS 2-5) / mild stroke (mRS 0,1) / TIA / no stroke-TIA, measured at 90 days.; this approach allows for smaller sample sizes compared to binary outcomes such as stroke/no stroke

SECONDARY OUTCOMES:
Safety | 90 days
  Days 7 and 35 Full blood count by local investigator
  Days 7, 35 and 90:
  Ordinal bleeding (fatal/major/moderate/minor/none42) as adjudicated by an independent blinded panel; death; binary major bleeding (fatal, symptomatic, causing fall in haemoglobin of ≥2g/l, or leading to transfusion of ≥2 units of blood/red cells);45 binary minor bleeding (e.g. bruising) binary bleeding; all bleeding, symptomatic intracerebral haemorrhage, major extracranial bleeding, binary serious adverse events, ordinal adverse events (fatal/serious/other/none42); thrombotic thrombocytopenic purpura; granulocytopenia.
Serious adverse events | 90 Days
Death | 90 days
Platelet function. | 90 Days
  Days 7 and 35 Full blood count by local investigator
  Days 7, 35 and 90:
  Ordinal bleeding (fatal/major/moderate/minor/none42) as adjudicated by an independent blinded panel; death; binary major bleeding (fatal, symptomatic, causing fall in haemoglobin of ≥2g/l, or leading to transfusion of ≥2 units of blood/red cells);45 binary minor bleeding (e.g. bruising) binary bleeding; all bleeding, symptomatic intracerebral haemorrhage, major extracranial bleeding, binary serious adverse events, ordinal adverse events (fatal/serious/other/none42); thrombotic thrombocytopenic purpura; granulocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bath, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: TARDIS Trial Website — http://www.tardistrial.org/